CLINICAL TRIAL: NCT01091662
Title: Double-Blind, Randomized, Historical Control Study of the Safety and Efficacy of Eslicarbazepine Acetate Monotherapy in Subjects With Partial Epilepsy Not Well Controlled by Current Antiepileptic Drugs
Brief Title: Safety & Efficacy of Eslicarbazepine Monotherapy in Sub.w/Partial Epilepsy Not Well Controlled by Current Antiepileptic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 093-046
Record Dates: First submitted 2010-03-17; First posted 2010-03-24 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-09

CONDITIONS: Epilepsy
Keywords: Seizures; Epilepsy; Anticonvulsant; Monotherapy; Historical control
MeSH Terms: conditions — Epilepsy; Seizures | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- eslicarbazepine acetate 1600 mg (Experimental): Subjects randomized to 1600 mg QD of eslicarbazepine acetate will titrate from 600 mg QD(Day 0) to 1200 mg once a day(Week 2) to 1600 mg QD (Weeks 3-18) and may taper down from 1600 mg to 800 mg QD 3 days after the Week 18 visit.
  Interventions: Drug: Eslicarbazepine acetate 1600 mg
- eslicarbazepine acetate 1200 mg (Experimental): Subjects randomized to 1200 mg QD eslicarbazepine acetate will titrate from 400 mg QD (Day0) to 800 mg QDweek2) to 1200 mg QD(weeks 3-18) and may taper down from 1200 mg to 600 mg QD 3 days after the Week 18 visit.
  Subjects may continue in an open-label extension study with a starting dose of 1200 mg QD, or taper off their previous antiepileptic drugs during weeks 2-8.
  Interventions: Drug: Eslicarbazepine acetate 1200 mg

INTERVENTIONS:
Drug: Eslicarbazepine acetate 1600 mg — 1600 mg once per day
  Arms: eslicarbazepine acetate 1600 mg
Drug: Eslicarbazepine acetate 1200 mg — 1200 once per day
  Arms: eslicarbazepine acetate 1200 mg

SUMMARY:
This is an 18-week, double-blind, multicenter study with gradual conversion from previous antiepileptic therapy to eslicarbazepine acetate monotherapy in subjects with partial epilepsy.

DETAILED DESCRIPTION:
This is an 18-week, double-blind, randomized, historical control, multicenter study with gradual conversion to monotherapy in subjects with partial onset seizures who are not well controlled by current AEDs. The 18 week double-blind treatment period consists of a 2-week titration period, 6-week taper or conversion period, and a 10-week monotherapy period. This study was previously posted by Sepracor Inc. In October 2009, Sepracor Inc. was acquired by Dainippon Sumitomo Pharma., and in October 2010, Sepracor Inc's name was changed to Sunovion Pharmaceuticals Inc.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of partial epilepsy as defined in the Classification of Seizures of the International League Against Epilepsy (ILAE) (simple partial seizures with observable motor component, or complex, with or without secondary generalization)

  * Medical history of seizures;
  * Absence of confounding factors (pseudoseizures, syncope);
  * Documented EEG recording (done within 5 years prior to screening) consistent with focal onset epilepsy
* Documented CT or MRI scan conducted within 10 years prior to screening, showing the absence of a structural abnormality (eg, tumor or malformation)
* ≥ 4 partial onset seizures during the 8 weeks prior screening with no 28-day seizure free period
* Stable treatment with 1-2 AEDs during the last 4 weeks prior to screening
* Subjects must have the ability to comprehend the informed consent form and be willing to provide informed consent. For subjects who are unable to comprehend the written consent, a witness/caregiver who is able to describe and provide an understanding of the informed consent to the subject must sign the consent form on behalf of the subject.
* Subjects must give written informed consent prior to participation in the study. For subjects <18 years of age, the informed consent must be signed by the subject's parent or legal guardian, and, when appropriate and/or required by state or local law, minor subjects must give written informed assent prior to participation in the study. Subjects of Asian ancestry are required to give written informed consent for genotyping. All subjects must sign a HIPAA Form. All females of child bearing potential must also sign the "Women of Childbearing Potential" Addendum.
* A female subject is eligible to enter and participate in the study if she is of:

  * Non-childbearing potential (ie, physiologically incapable of becoming pregnant, including any female who is pre-menarchal or post-menopausal);
  * Child-bearing potential (all females ≤65 years of age), has a negative pregnancy test at screening and agrees to satisfy contraception requirements

Exclusion Criteria:

* Subjects with only simple partial seizures without a motor component
* Presence of generalized seizure syndromes (eg, juvenile myoclonic epilepsy or Lennox-Gastaut syndrome)
* History of pseudo-seizures
* Current seizures related to an acute medical illness
* Seizures secondary to metabolic, toxic or infectious disorder or drug abuse
* Status epilepticus within 2 years prior to screening
* Seizures only occurring in a cluster pattern
* Subjects taking 2 of the following sodium channel blocking AEDs: phenytoin, carbamazepine, oxcarbazepine, or lamotrigine
* Subjects taking 2 AEDs with both being in the upper dose range (defined as approximately two-thirds of the defined daily dose)
* Subjects taking more than 2 AEDs
* Subjects with progressive structural central nervous system lesion or progressive encephalopathy
* Psychiatric exclusion criteria
* Medical exclusion criteria: known renal insufficiency (estimated creatinine clearance [CrCL]) <60 mL/min based on serum creatinine using the Cockcroft-Gault formula
* Clinical and laboratory exclusion criteria: Subjects of Asian ancestry who tests positive for the presence of the HLA-B*1502 allele
* Subjects who have been on benzodiazepines, phenobarbital, or primidone on a regular basis within 3 months prior to screening
* Subjects taking antipsychotics, tricyclic antidepressants, anxiolytics, sedative hypnotics including non-benzodiazepines, central opioid agonists/antagonists, monoamine oxidase inhibitors (MAOIs) within at least 5 half lives (or for at least 2 weeks whichever is longer) prior to randomization
* Subjects presently on felbamate or vigabatrin

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Dirctor, Study Director — Sumitomo Pharma America, Inc.
Locations (62):
- United States (39):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Neurology, Conway, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kern County Neurological Medical Group, INC., Bakersfield, California
  - Neuro-Pain Medical Center, Fresno, California
  - West Los Angeles VA Medical Center, Los Angeles, California
  - Neurosearch II Inc., Ventura, California
  - Specialty Nuerology, PC, Englewood, Colorado
  - Palm Springs Research Institute, Inc, Hialeah, Florida
  - Miami Children's Hospital, Miami, Florida
  - Pharma Care Research LLC, Miami, Florida
  - Bay Neurological Institute, Panama City, Florida
  - Loveland Scientific Resources Inc., Venice, Florida
  - Josephson Wallack Munshower Neurology PC, Indianapolis, Indiana
  - University of Kentucky Department of Neurology, Lexington, Kentucky
  - Louisiana State University Health Science Center - Shreveport, Shreveport, Louisiana
  - The Sandra and Malcom Berman Brain & Spine Institute, Baltimore, Maryland
  - Lahey Clinic, Burlington, Massachusetts
  - Wayne State University/Detroit Medical Center, Detroit, Michigan
  - Minneappolis Clinic of Neurology, Golden Valley, Minnesota
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - UMDNJ DOC 8th Floor 8100, Newark, New Jersey
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - Shore Neurology, PA, Toms River, New Jersey
  - Dent Neurologic Institute, Orchard Park, New York
  - SUNY Upstate Medical University Department of Neurology, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - East Carolina Neurology, Greenville, North Carolina
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Tulsa Clinical Research LLC, Tulsa, Oklahoma
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Community Clinical Research Inc., Austin, Texas
  - Brownwood Regional Medical Center, Brownwood, Texas
  - MD, Dallas, Texas
  - Vital Clinical Research, DeSoto, Texas
  - Marshfield Clinic, Marshfield, Wisconsin
  - Regional Epilepsy Center, Milwaukee, Wisconsin
- Bulgaria (4):
  - Multirprofile Hospital for Active Treatment "Pulse," AD, town of Blagoevgrad, Blagoevgrad, Bulgaria
  - Second Multiprofile Hospital for Active Treatment - Sofia, AD, city of Sofia Neurology Department, Sofia, Bulgaria
  - University Multiprofile Hospital for Active Treatment "Dr. Georgi Stranski," EAD, town of Pleven, Pleven, Pleven
  - Diagnostic and Consultative Center "Equita" EOOD, town of Varna, Varna, Varna
- Czechia (6):
  - Policlinic Chocen, private neurology, Smetanova, Chocen
  - Prague, Pocernicka
  - Neurologicka ordinance, Kolejni, Prague
  - CTC Rycnov nad Kneznou, Rychnov nad Kněžnou, Praugue
  - Cerebrovaskularni poradna s.r.o., Ostrava, Tiebovice
  - Poradna pro epilepsie, Koterova, Zin
- Serbia (2):
  - Clinic of Neurology, Clinical Center of Serbia, Belgrade, Belgrade
  - Institute of Mental Health, Department of epilepsy and clinical neurophysiology, Palmoticeva, Belgrade
- Ukraine (11):
  - Communal Institution "Dnipropetrovsk Regional Clinical Hospital named after l.l. Mechnikov" Regional Center of psychosomatic disorders, Psychoneurology department for patients with psychosomatic disorders and borderline condtions, Dnipropetrovsk, Dnipropetrovsk Oblast
  - Communal Medical and Preventive Treatment Institution "Regional Clincal Psychiatric Hospital" Donetsk National Medical University, Donetsk, Donetsk Oblast
  - State Institution "Institute of neurology, psychiatry and narcology of AMS of Ukraine" Department of cerebrovascular patology, Kharkiv, Kharkivs’ka Oblast’
  - State Treatment and Prevention Institution, Kharkiv, Kharkov
  - State Institution "Institute of the Health Care of Children & Adolescents of Academy of Medical Sciences of Ukraine" Dept of Psychiatry, Kharkiv, Kharkov
  - State Institution Railway Clinical Hospital #1 of Kiev Railway Station of DTGO South Western Railroad Psycho-neurological Department, Kiev, Kyiv City
  - Communal Institution "Lviv Regional Clinical Psychiatric Hospital" Department #20, Lviv National Medical University, named after Danylo, Lviv, Lviv Oblast
  - Communal Institution "Odessa Regional Clinical Psych Hospital #1" Department of Day Care, Odesa, Odesa Oblast
  - Poltava Regional Clinical Psychiatric Hospital named O.F. Maltsev, Poltava, Poltava Oblast
  - Crimean Republic Institution "Clinical Psychiatric Hospital #1", Simferopol, Simferopol
  - Communal Institution "Vinnytsia Regional Psycho-Neurological Hospital named after O.I. Yuschenko, Vinnytsia National Medical University named after M.I. Pirogov, Dispensary department, Department of Psychiatry and Addictology, Vinnytsia, Vinnytsia Oblast

REFERENCES:
- [Background] Jacobson MP, Pazdera L, Bhatia P, Grinnell T, Cheng H, Blum D; study 046 team. Efficacy and safety of conversion to monotherapy with eslicarbazepine acetate in adults with uncontrolled partial-onset seizures: a historical-control phase III study. BMC Neurol. 2015 Mar 28;15:46. doi: 10.1186/s12883-015-0305-5. PMID 25880756

RESULTS

PARTICIPANT FLOW:
Groups:
- ESL 1200 mg: Subjects randomized to 1200 mg QD eslicarbazepine acetate will titrate from 400 mg (Week 1) to 800 mg (Week 2) to 1200 mg (Weeks 3-18) QD and taper down from 1200 mg to 600 mg QD 3 days after the end of Week 18..
- ESL1600 mg: Subjects randomized to 1600 mg QD of eslicarbazepine acetate will titrate from 600 mg (Week 1) to 1200 mg (Week 2) to 1600 mg (Weeks 3-18) QD and taper down from 1600 mg to 800 mg QD 3 days after the end of Week 18.
Period: Overall Study
Arm/Group | ESL 1200 mg | ESL1600 mg
Started | 58 | 114
Completed | 41 | 80
Not Completed | 17 | 34
Not completed — Adverse Event | 1 | 9
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 7 | 6
Not completed — met exit criteria | 7 | 13
Not completed — met exclusion criteria | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — unable to swallow capsule | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- ESL1200 mg: Subjects randomized to 1200 mg QD eslicarbazepine acetate will titrate from 400 mg (Week 1) to 800 mg (Week 2) to 1200 mg (Weeks 3-18) QD and taper down from 1200 mg to 600 mg QD 3 days after the end of Week 18..
- ESL 1600 mg: Subjects randomized to 1600 mg QD of eslicarbazepineacetate will titrate from 600 mg (Week 1) to 1200 mg (Week 2) to 1600 mg (Weeks 3-18) QD and taper down from 1600 mg to 800 mg QD 3 days after the end of Week 18.
- Total: Total of all reporting groups
Arm/Group | ESL1200 mg | ESL 1600 mg | Total
Number analyzed (Participants) | 58 | 114 | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 4 | 7
  Between 18 and 65 years | 55 | 110 | 165
  >=65 years | 0 | 0 | 0
Age, Customized [Number; unit: participants]
  <18 years | 3 | 4 | 7
  18-39 years | 32 | 59 | 91
  40-65 years | 23 | 51 | 74
  >65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 62 | 89
  Male | 31 | 52 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 7 | 8
  Not Hispanic or Latino | 57 | 107 | 164
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Czech Republic | 11 | 22 | 33
  United States | 15 | 28 | 43
  Ukraine | 26 | 42 | 68
  Bulgaria | 6 | 19 | 25
  Serbia | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Cumulative 112-day Exit Rate as Estimated by Kaplan-Meier Method
Description: Cumulative exit rate was defined as the proportion of subjects meeting at least one of the following five exit criteria over a 16-week study period (from start of AED taper/con. period (Wk 3) to end of double blind monotherapy period (Wk 18)).1.One episode of status epilepticus.2.One secondary gen. partial seizure (in subjects who did not have gen.seizures during 6 mo. prior to screening).3.A two fold increase in any consecutive 28 day seizure rate compared to the highest consecutive 28 day seizure rate during the 8 week baseline period. 4.A two fold increase in any consecutive 2 day seizure rate compared to the highest consecutive 2 day seizure rate during the 8 week baseline period. If the highest number of seizures in any consecutive 2 day period during the 8 week baseline was 1 then 3 seizures in a consecutive 2 day period was required to exit.
  5.Worsening of seizures or increase in seizure frequency considered serious or requiring intervention as judged by the investigator
Time Frame: From beginning of Week 3 to end of Week 18
Population: Efficacy population
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- ESL1200 mg: Titrate from 400 mg (Week 1) to 800 mg (Week 2) to 1200 mg (Weeks 3-18) QD and taper down from 1200 mg to 600 mg QD 3 days after the end of Week 18.
- ESL 1600 mg: Titrate from 600 mg (Week 1) to 1200 mg (Week 2) to 1600 mg (Weeks 3-18) QD and taper down from 1600 mg to 800 mg QD 3 days after the end of Week 18.
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
proportion of participants | 0.156 [0.0810 to 0.2874] | 0.128 [0.0750 to 0.2152]

2. Secondary Outcome: Proportion (%) of Subjects That Are Seizure-free During the 10-week Double-blind Monotherapy Treatment Period.
Description: Seizure-free subjects during the monotherapy period were determined as subjects who had seizure assessments during the monotherapy period, and did not have any seizures in the 10 weeks between Visits 6 and 9 (Weeks 9 through 18). Subjects who discontinued during this period were considered not seizure-free even if they were seizure-free at the time of discontinuation, i.e., to be considered seizure-free, subjects must complete the 10-week period without any seizures.
Time Frame: Week 9 through 18
Population: Efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
percentage of participants | 7.4 [2.1 to 17.9] | 10.0 [4.9 to 17.6]

3. Secondary Outcome: Percentage of Subjects Seizure-free During the Last 4 Weeks on Eslicarbazepine Acetate Monotherapy.
Description: Percentage of participants that were Seizure-free during the last four weeks of monotherapy were determined as subjects who had seizure assessments during the 4 weeks between Visits 8 and 9 (Weeks 15 through 18), and did not have any seizures.
Time Frame: Week 15 through 18
Population: Efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
percentage of participants | 16.7 [7.9 to 29.3] | 17.0 [10.2 to 25.8]

4. Secondary Outcome: Completion Rate (% of Subjects Completing the 18 Weeks of Double-blind Treatment).
Description: Subjects completing the study were determined as subjects who completed the 18 weeks of double-blind treatment.
Time Frame: 18 weeks
Population: Efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
percentage of participants | 75.9 [62.4 to 86.5] | 80.0 [70.8 to 87.3]

5. Secondary Outcome: Completion Rate During the 10 Weeks of Monotherapy (% of Subjects Entering the Monotherapy Period Who Complete).
Description: Monotherapy completion rate was defined as the proportion (%) of subjects entering the monotherapy period who completed the 10 weeks of monotherapy treatment.
Time Frame: Week 8 through 18
Population: Efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
percentage of participants | 85.4 [72.2 to 93.9] | 90.9 [82.9 to 96.0]

6. Secondary Outcome: Time on Eslicarbazepine Acetate Monotherapy.
Description: The start of the monotherapy period was defined as the date of termination of all other AEDs while taking study monotherapy medication. Time on monotherapy was defined from the start of monotherapy period to the last dose of monotherapy treatment.
Time Frame: Week 8 to Week 18
Population: Efficacy population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
days | NA [NA to NA] — median not calculable due to lack of events | NA [NA to NA] — median not calculable due to lack of events

7. Secondary Outcome: Change in Seizure Frequency From Baseline.
Description: The relative (%) change in standardized seizure frequency was evaluated for four periods: titration (Weeks 1 to 2), AED taper/conversion (Weeks 3 to 8), monotherapy (Weeks 9 to 18), and double-blind (Weeks 1 to 18).
Time Frame: 18 weeks, Double-blind:weeks 1-18; Baseline: weeks -8to -1; titration: weeks 1 to 2; AED taper/conversion: weeks 3 to 8; monotherapy; weeks 9 to 18
Population: Efficacy population (ESL 1200mg) Double-blind: 54; Titration: 54; AED taper/conversion:54; Monotherapy: 48 (ESL1600 mg) Double-blind:98; Titration: 98; AED taper/conversion: 98; Monotherapy: 87
Measure: Median (Inter-Quartile Range); unit: Percent change
Groups:
- ESL 1200 mg: Titrate from 400 mg (Week 1) to 800 mg (Week2) to 1200 mg (Weeks 3-18) QD and taper down from 1200 mg to 600 mg QD 3 days after end of Week 18.
- ESL 1600 mg: Titrate from 600 mg (Week 1) to 1200 mg (Week 2) to 1600 mg (Weeks 3-18) QD and taper down from 1600 mg to 800 mg QD 3 days after end of Week 18.
Arm/Group | ESL 1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 98
Percent change
  Relative(%) change from baseline fo DB pd n=54,98 | -36.1 [-59.2 to -17.1] | -47.5 [-70.8 to -11.3]
  Relative(%)chg from baseline for titrat pd n=54,98 | -19.3 [-57.9 to 3.3] | -35.6 [-72.4 to -9.4]
  Relative (%) chg from baseline-AED t/c pd n=54,98 | -39.4 [-54.0 to 0.0] | -42.9 [-73.8 to -12.1]
  Relative (%) change from baseline-mono pd n=48,87 | -45.7 [-72.1 to -20.1] | -52.1 [-81.6 to -21.8]

8. Secondary Outcome: Responder Rate (Proportion [%] of Subjects With a ≥50% Reduction of Seizure Frequency From Baseline).
Description: Responder rate was defined as the proportion (%) of subjects with a ≥ 50% reduction of seizure frequency from baseline. This analysis was done for the titration (Weeks 1 to 2), AED taper/conversion (Weeks 3 to 8), monotherapy (Weeks 9 to 18), and double-blind (Weeks 1 to 18) periods.
Time Frame: Week 0 to Week 18, Double-blind weeks 1-18; baseline: weeks -8 to -1; Titration: weeks 1-2; AED taper/conversion; weeks 3-8; monotherapy weeks 9-18
Population: Efficacy population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ESL1200 mg: Titrate from 400 mg (Week 1) to 800 mg (Week2) to 1200 mg (Weeks 3-18) QD and taper down from 1200 mg to 600 mg QD 3 days after end of Week 18.
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
percentage of participants
  responder rate during the DB period | 35.2 [22.7 to 49.4] | 46.0 [36.0 to 56.3]
  responder rate during titration period | 29.6 [18.0 to 43.6] | 37.0 [27.6 to 47.2]
  responder rate during the AED | 29.6 [18.0 to 43.6] | 39.0 [29.4 to 49.3]
  responder rate during monotherapy period | 38.9 [29.5 to 58.8] | 46.0 [41.4 to 63.0]

9. Secondary Outcome: Proportion (%) of Subjects Reaching Each Exit Criteria
Description: The proportion (%) of subjects reaching each of the 5 exit criteria-1.One episode of status epilepticus.2.One secondary gen. partial seizure (in subjects who did not have gen.seizures during 6 mo. prior to screening).3.A two fold increase in any consecutive 28 day seizure rate compared to the highest consecutive 28 day seizure rate during the 8 week baseline period. 4.A two fold increase in any consecutive 2 day seizure rate compared to the highest consecutive 2 day seizure rate during the 8 week baseline period. If the highest number of seizures in any consecutive 2 day period during the 8 week baseline was 1 then 3 seizures in a consecutive 2 day period was required to exit.
  5.Worsening of seizures or increase in seizure frequency considered serious or requiring intervention as judged by the investigator
Time Frame: Week 1 to Week 18, (beginning of week 1 to end of week 18)
Population: Efficacy population
Measure: Number; unit: percentage of participants
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
percentage of participants
  exit criterion 1 | 0 | 0
  exit criterion 2 | 1.9 | 0
  exit criterion investigator prog. assessment) | 5.6 | 2.0
  exit criterion 3 (sponsors prog. assessment) | 3.7 | 1.0
  exit criterion 4 (investigaor prog. assessment) | 1.9 | 5.0
  exit criterion 4 (sponsor prog. assessment) | 3.7 | 6.0
  exit criterion 5 | 3.7 | 5.0

10. Secondary Outcome: Change in Total Score From Baseline in 31-Item Quality of Life in Epilepsy (QOLIE-31).
Description: The QOLIE-31 overall score was obtained by using a weighted average of multi-item scale scores. The recorded responses were converted to 0-100 point scales. The mean of the individual item scores in each subgroup were calculated, with higher converted scores reflecting better quality of life.
Time Frame: Week 0 to Week 18, Baseline: Day 0: End of AED taper/conversion period: end of week 8; End of monotherapy period: end of week 18
Population: Efficacy Population (ESL 1200 mg) Change from baseline to end of AED taper/conversion period: 45; Change from baseline to end of monotherapy period:50 (ESL1600 mg) Change from baseline to end of AED taper/conversion period: 85; Change from baseline to end of monotherapy period:96
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 50 | 96
units on a scale
  chg from baseline-end of AED taper/covn.pd n=45,85 | 3.4 (12.03) | 5.8 (11.77)
  change from baseline-end of monotherapy pd n=50,96 | 4.0 (11.48) | 4.7 (13.70)

11. Secondary Outcome: Change in Total Score in Montgomery-Asberg Depression Rating Scale (MADRS),From Baseline .
Description: The total score of MADRS is defined as the sum of all individual item scores. From 0-60, high score indicates more severe
Time Frame: Week 0 to Week 18,baseline day 0; end of AED taper/conversion period; end of week 8; end of monotherapy period; end of week 18
Population: Efficacy Population (ESL 1200 mg) Change from baseline to end of AED taper/conversion period: 48; Change from baseline to end of monotherapy period: 54 (ESL 1600 mg) Change from baseline to end of AED taper/conversion period: 88; Change from baseline to end of monotherapy period: 98
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
units on a scale
  chg from baseline-end of AED taper/covn.pd n=48,88 | -1.2 (3.69) | -1.8 (4.01)
  chg from baseline-end of monotherapy pd n=54,98 | 0.0 (6.47) | -1.6 (4.54)

12. Secondary Outcome: Change in Total Score of MADRS From Baseline in Those Subjects With a MADRS Score of ≥14 at Randomization.
Description: The total score of MADRS is defined as the sum of all individual item scores. From 0-60, higher score indicates more severe
Time Frame: Week 0 to Week 18, baseline:day 0;end of AED taper/conversion period; end of week 8; end of monotherapy period: end of week 18
Population: efficacy population (ESL 1200 mg) Change from baseline to end of AED taper/conversion period: 7; Change from baseline to end of monotherapy period: 7 (ESL 1600 mg) Change from baseline to end of AED taper/conversion period: 16; Change from baseline to end of monotherapy period: 18
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 50 | 100
units on a scale
  chge from baseline-end of AED taper/covn.pd n=7,16 | -3.9 (4.30) | -6.6 (4.15)
  chg from baseline-end of monotherapy pd n=7,18 | -6.1 (6.72) | -4.1 (7.58)

13. Secondary Outcome: Proportion (%) of Subjects With Increase of Body Weight >= 7% From Baseline
Time Frame: 18 Week Double-blind treatment period
Population: ITT population
Measure: Number; unit: percentage of participants
Groups:
- ESL 1600 mg: Subjects randomized to 1600 mg QD of eslicarbazepine acetate will titrate from 600 mg (Week 1) to 1200 mg (Week 2) to 1600 mg (Weeks 3-18) QD and taper down from 1600 mg to 800 mg QD 3 days after the end of Week 18.
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 58 | 114
percentage of participants | 1.8 | 11.7

14. Secondary Outcome: Proportion (%) of Subjects With Normal Baseline Sodium Reaching Blood Sodium ≤135 mmol/L, ≤130 mmol/L, and ≤125 mmol/L.
Description: Proportion (%) of Subjects With Normal Baseline Sodium Reaching Blood Sodium ≤135 mmol/L, ≤130 mmol/L, and ≤125 mmol/L
Time Frame: Week 0 to Week 18
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 58 | 114
percentage of participants
  ≤ 135 and > 130 mEq/L | 49.1 | 54.5
  ≤ 130 and > 125 mEq/L | 8.8 | 20.9
  ≤ 125 mEq/L | 0 | 0

15. Secondary Outcome: Proportion (%) of Events in Each Classification of the Columbia Suicide Severity Rating Scale (C SSRS).
Time Frame: 18 Week Double-blind treatment period
Population: ITT population
Measure: Number; unit: Percent of particiants
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 58 | 114
Percent of particiants
  Actual Attempt | 3.4 | 0
  Non-suicidal Self-Injurious Behavior | 0 | 0.9
  Interrupted Attempt | 0 | 0
  Aborted Attempt | 0 | 0
  Preparatory Attempts | 0 | 0
  Suicidal Behavior | 3.4 | 0
  Wish to be Dead | 1.7 | 0.9
  Non-specific Active Suicidal Thoughts | 0 | 1
  Act. Suicidal Idea. w/any method-no intent to act | 0 | 0
  Act. Suicidal Idea.w/any method-some intent to act | 0 | 0.9
  Act. Suicidal Idea. w/any method-Spec. Plan to act | 0 | 0

16. Secondary Outcome: Standardized Seizure Frequency (SSF) by Period
Description: Seizure frequency was evaluated by using a standardized frequency per 4 weeks (28 days). It was evaluated for five periods: baseline (Weeks -8 to -1), titration (Weeks 1 to 2), AED taper/conversion (Weeks 3 to 8), monotherapy (Weeks 9 to 18), and double-blind (Weeks 1 to 18).
Time Frame: Double-blind: week to 18; Baseline: weeks -8 to -1; titration: weeks 1 to 2; AED taper/conversion weeks 3 to 8; monotherapy: weeks 9 to 18
Population: efficacy population (ESL 1200 mg) Double-blind: 54; Baseline: 54; Titration: 54; AED taper/conversion; 54; Monotherapy: 48 (ESL 1600 mg) Double-blind: 100; Baseline: 98; Titration: 100; AED taper/conversion; 100; Monotherapy: 88
Measure: Mean (Standard Deviation); unit: seizures in 28 days
Arm/Group | ESL1200 mg | ESL 1600 mg
Number analyzed (Participants) | 54 | 100
seizures in 28 days
  SSF during double-blind pd n=54,100 | 5.5 (7.75) | 5.2 (5.38)
  SSF druing baseline pd n=54,98 | 7.4 (5.89) | 8.7 (7.20)
  SSF during titration pd n=54,100 | 6.0 (6.16) | 6.4 (8.11)
  SSF during AED taper/conversion pd n=54,100 | 6.0 (9.68) | 5.1 (5.26)
  SSF during monotherapy pd n=48,88 | 4.7 (6.10) | 5.0 (5.62)

ADVERSE EVENTS:
Time Frame: 18 week double-blind treatment period
Arm/Group | ESL1200 mg | ESL 1600 mg
Serious Adverse Events (participants affected / at risk) | 1/58 | 8/114
Other Adverse Events (participants affected / at risk) | 29/58 | 64/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESL1200 mg (N=58) | ESL 1600 mg (N=114)
Atrial flutter (Cardiac disorders) | 1 (1) | 1 (1)
ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Complex partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Partial seizures with secondary generalisation (Nervous system disorders) | 0 (0) | 1 (1)
Synocope (Nervous system disorders) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Drug rash with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESL1200 mg (N=58) | ESL 1600 mg (N=114)
Nausea (Gastrointestinal disorders) | 6 (8) | 7 (12)
Fatigue (General disorders) | 4 (5) | 6 (7)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 9 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (7)
Dizziness (Nervous system disorders) | 6 (7) | 24 (37)
Headache (Nervous system disorders) | 11 (16) | 32 (87)
Solmnolence (Nervous system disorders) | 2 (2) | 10 (12)
Anxiety (Psychiatric disorders) | 3 (4) | 1 (1)
Insomnia (Psychiatric disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.